CLINICAL TRIAL: NCT00458432
Title: Functional Neuroanatomy of Emotion Perception, Recognition, Learning, and Memory
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070127; 07-M-0127
Record Dates: First submitted 2007-04-07; First posted 2007-04-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-08

CONDITIONS: Healthy
Keywords: fMRI; Pavlovian Conditioning; Functional Activity; Brain; Fear; Healthy Volunteer; HV

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study uses magnetic resonance imaging (MRI) to explore the areas of the brain involved in different types of mental processes, in particular, the brain regions involved in perception, recognition, learning, and memory. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. In this study it is also used to measure blood flow in different regions of the brain while the subject is presented auditory or visual stimuli. The subject lies on a table that can slide in and out of the scanner (a narrow cylinder), wearing earplugs to muffle loud noises that occur during the scanning process. Subjects are in the scanner no more than 2 hours.

Healthy, right-handed normal volunteers between 20 and 40 years of age who have at least a high school education may be eligible for this study.

While undergoing MRI, participants are presented visual stimuli (pictures or geometric shapes on a projection screen) or auditory stimuli (tones played through a set of headphones). Unpleasant stimuli such as loud noise, electric shocks, heat, or tactile stimuli are administered occasionally. The intensity of these stimuli is similar to those experienced in practice sessions before the scanning. Participants receive between 30 and 60 visual or auditory stimuli during the scanning session, and each stimulus lasts about 1 second. In some studies participants are asked to move a joystick that controls a rating bar presented on a projection screen to indicate when they expect to receive these stimuli and how sure they are that they will occur. Heart rate, respiration rate, and sweat gland activity are monitored during the MRI sessions, using electrodes placed on the fingers to measure heart rate and sweat gland activity and a sensor strapped around the chest to measure respiration. Subjects are in the scanner no more than 2 hours.

Following the experiment, subjects may be asked questions about their experiences during the study.

DETAILED DESCRIPTION:
The long-term goals of this study are to understand the neural substrates of aversive Pavlovian conditioning in human subjects. The general approach is to use whole brain functional magnetic resonance imaging (fMRI) to describe brain regions and circuits that contribute to the acquisition and performance of this form of learning. The specific aims of this proposal are:

1. To identify brain regions that respond to aversive stimuli.
2. To identify brain regions primarily responsible for the expression of cognitive and autonomic responses versus those involved in stimulus processing and memory encoding.
3. To relate patterns of activity within selected brain areas to implicit versus explicit memory performance.
4. To compare the parallel development of implicit and explicit knowledge about stimulus relationships during Pavlovian delay and trace fear conditioning.
5. To test specific predictions regarding the nature of learning-related activity in the amygdala, hippocampus, anterior cingulate, and prefrontal cortex as they develop during conditioning and to integrate these findings into a more general theoretical understanding of memory phenomena in humans.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal right-handed volunteers with at least a high school education, age 20 to 40 years, will be recruited to participate in this study.

EXCLUSION CRITERIA:

Subjects will be excluded if they have evidence of or a history of learning disability, psychiatric condition, head trauma, seizures or other neurological condition, alcoholism or substance abuse, hypertension, or cardiovascular disease. We will also exclude subjects with vision and/or hearing problems severe enough to interfere with testing. Lab work will be limited to a urine pregnancy test for females. Females with a positive pregnancy test will be excluded from neuroimaging studies. All subjects will be questioned prior to MRI scanning for possible occupational exposure to metal slivers or shavings, which may have become accidentally lodged in the tissues of the head or neck. Those whose history is suggestive of such a problem will be excluded. Subjects with surgical clips or shrapnel in or near the brain or blood vessels, subjects with cochlear implants, subjects with any metallic body in the eye or CNS, and subjects with any form of implant wire or metal device which may concentrate radiofrequency fields will be excluded because of possible risks during MRI scanning.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180
Dates: Start 2007-04-05; Primary Completion 2009-08-31 (Actual); Study Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baumgartner U, Magerl W, Klein T, Hopf HC, Treede RD. Neurogenic hyperalgesia versus painful hypoalgesia: two distinct mechanisms of neuropathic pain. Pain. 2002 Mar;96(1-2):141-51. doi: 10.1016/s0304-3959(01)00438-9. PMID 11932070
- [Background] Bechara A, Tranel D, Damasio H, Adolphs R, Rockland C, Damasio AR. Double dissociation of conditioning and declarative knowledge relative to the amygdala and hippocampus in humans. Science. 1995 Aug 25;269(5227):1115-8. doi: 10.1126/science.7652558.
- [Background] Andrew D, Greenspan JD. Peripheral coding of tonic mechanical cutaneous pain: comparison of nociceptor activity in rat and human psychophysics. J Neurophysiol. 1999 Nov;82(5):2641-8. doi: 10.1152/jn.1999.82.5.2641. PMID 10561433